CLINICAL TRIAL: NCT00721955
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Multi-Dose Efficacy and Safety Study of Staccato® Loxapine for Inhalation in Patients With Bipolar I Disorder and Acute Agitation
Brief Title: Staccato Loxapine in Agitated Patients With Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-004-302
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2008-10

CONDITIONS: Bipolar I Disorder
Keywords: Bipolar 1 disorder,; agitation,; acute,; treatment
MeSH Terms: conditions — Psychomotor Agitation | interventions — Loxapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Inhaled Placebo (Placebo Comparator): Inhaled Staccato Placebo, may repeat after 2 hours x 2
  Interventions: Drug: Inhaled Placebo
- Inhaled Loxapine 5 mg (Experimental): Inhaled Staccato Loxapine 5 mg, may repeat after 2 hours x 2
  Interventions: Drug: Inhaled loxapine 5 mg
- Inhaled Loxapine 10 mg (Experimental): Inhaled Staccato Loxapine 10 mg, may repeat after 2 hours x 2
  Interventions: Drug: Inhaled loxapine 10 mg

INTERVENTIONS:
Drug: Inhaled Placebo — Inhaled loxapine Placebo, may repeat after 2 hours x 2
  Other Names: Staccato Placebo
  Arms: Inhaled Placebo
Drug: Inhaled loxapine 5 mg — Inhaled Staccato loxapine 5 mg, may repeat after 2 hours x 2
  Other Names: ADASUVE 5 mg
  Arms: Inhaled Loxapine 5 mg
Drug: Inhaled loxapine 10 mg — Inhaled Staccato loxapine 10 mg, may repeat after 2 hours x 2
  Other Names: ADASUVE 10 mg
  Arms: Inhaled Loxapine 10 mg

SUMMARY:
Phase 3 safety and efficacy study of Staccato Loxapine in the treatment of acute agitation in bipolar 1 disorder patients.

DETAILED DESCRIPTION:
This is an in-clinic, multi-center, randomized, double-blind, placebo-controlled study of 2 dose levels of Staccato Loxapine, 5 and 10 mg. Patients may receive up to 3 doses of study drug in a 24-hour period, depending on their clinical status. The primary endpoint is the change from baseline in the PANSS (Positive and Negative Symptom Scale) Excited Component (also known as PEC) score, performed at 2 hours after the first dose.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients with bipolar 1 disorder and acute agitation

Exclusion Criteria:

* Agitation caused primarily by acute intoxication
* History of drug or alcohol dependence
* Treatment with benzodiazepines or other hypnotics within 4 hours prior to study drug administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Fishman, MD, Study Director — Alexza Pharmaceuticals, Inc.
Locations (6):
- United States (6):
  - Synergy Escondido, Escondido, California
  - Collaborative NeuroScience Network, Inc., Garden Grove, California
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - FutureSearch Trials, Austin, Texas
  - Claghorn-Lesem Research Clinic, Houston, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

REFERENCES:
- [Background] Kwentus J, Riesenberg RA, Marandi M, Manning RA, Allen MH, Fishman RS, Spyker DA, Kehne JH, Cassella JV. Rapid acute treatment of agitation in patients with bipolar I disorder: a multicenter, randomized, placebo-controlled clinical trial with inhaled loxapine. Bipolar Disord. 2012 Feb;14(1):31-40. doi: 10.1111/j.1399-5618.2011.00975.x. PMID 22329470
- [Derived] Zeller S, Zun L, Cassella JV, Spyker DA, Yeung PP. Response to inhaled loxapine in patients with schizophrenia or bipolar I disorder: PANSS-EC responder analyses. BJPsych Open. 2017 Nov 10;3(6):285-290. doi: 10.1192/bjpo.bp.117.005363. eCollection 2017 Nov. PMID 29163985

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg
Started | 105 | 104 | 105
Completed | 105 | 104 | 103
Not Completed | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg | Total
Number analyzed (Participants) | 105 | 104 | 105 | 314
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 105 | 104 | 105 | 314
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (9.82) | 41.2 (9.63) | 40.5 (9.80) | 40.7 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 57 | 52 | 158
  Male | 56 | 47 | 53 | 156
Region of Enrollment [Number; unit: participants]
  United States | 105 | 104 | 105 | 314

OUTCOME MEASURES:

1. Primary Outcome: Change in PANSS Excited Component (PEC) Score From Baseline Following Dose #1 of Staccato Loxapine, Compared With Placebo
Description: The Positive and Negative Syndrome Scale-Excited Component (PANSS-EC) comprises 5 items associated with agitation: poor impulse control, tension, hostility, uncooperativeness, and excitement; each scored 1 (min) to 7 (max). The PANSS-EC, the sum of these 5 subscales, thus ranges from 5 to 35. Individuals were eligible if they had a PANSS-EC of ≥14 (out of 35) and a score ≥4 (out of 7) on at least 1 of the 5 items.
Time Frame: Baseline and 2 hours
Population: ITT Population with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg
Number analyzed (Participants) | 105 | 104 | 105
units on a scale | -4.9 (4.77) | -8.1 (4.90) | -9.0 (4.67)
Statistical Analysis 1: Comparison: Inhaled Placebo vs Inhaled Loxapine 5 mg; Test type: Superiority — LS mean was used in the primary efficacy analysis; p < 0.0001, ANCOVA — p-values (adjusted) using Dunnett's t-test in main effects ANCOVA model
Statistical Analysis 2: Comparison: Inhaled Placebo vs Inhaled Loxapine 10 mg; Test type: Superiority — p-values (adjusted) using Dunnett's t-test in main effects ANCOVA model; p < 0.0001, ANCOVA — p-values (adjusted) using Dunnett's t-test in main effects ANCOVA model

2. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Score Following Dose #1 of Staccato Loxapine, Compared With Placebo
Description: Clinical Global Impression- Improvement (CGI-I) scores ranged from 1 to 7: 0=not assessed (missing), 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse.
Time Frame: Baseline and 2 hours
Population: ITT Population with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg
Number analyzed (Participants) | 105 | 104 | 105
units on a scale | 3.0 (0.99) | 2.1 (1.10) | 1.9 (1.14)
Statistical Analysis 1: Comparison: Inhaled Placebo vs Inhaled Loxapine 5 mg; Test type: Superiority — LS mean was used in the primary efficacy analysis; p < 0.0001, ANCOVA — p-values (adjusted) using Dunnett's t-test in main effects ANCOVA model
Statistical Analysis 2: Comparison: Inhaled Placebo vs Inhaled Loxapine 10 mg; Test type: Superiority; p < 0.0001, ANCOVA — -values (adjusted) using Dunnett's t-test in main effects ANCOVA model

3. Secondary Outcome: CGI-I Responders
Description: Frequency of response based on the CGI-I (defined as achieving a CGI-I score of 1 or 2 at 2 hours after administration of the inhalation)
Time Frame: Baseline and 2 hours
Population: ITT Population with LOCF
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg
Number analyzed (Participants) | 105 | 104 | 105
Participants | 29 | 69 | 78

ADVERSE EVENTS:
Time Frame: From informed consent through 30 days after last treatment
Description: AEs were recorded when identified by the study center staff or volunteered by a patient.
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/104 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/104 | 0/105
Other Adverse Events (participants affected / at risk) | 26/105 | 35/104 | 31/105
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Placebo (N=105) | Inhaled Loxapine 5 mg (N=104) | Inhaled Loxapine 10 mg (N=105)
Dysgeusia (Gastrointestinal disorders) | 6 (6) | 18 (18) | 18 (18)
Dizziness (Nervous system disorders) | 8 (8) | 6 (6) | 5 (5)
Headache (Musculoskeletal and connective tissue disorders) | 9 (9) | 4 (4) | 2 (2)
Sedation (Nervous system disorders) | 3 (3) | 7 (7) | 6 (6)

LIMITATIONS AND CAVEATS:
Because of the need to provide informed consent, the types of patients enrolled in the study may not have been representative of the most severely agitated patients who present for emergency care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less